CLINICAL TRIAL: NCT04071158
Title: A PHASE 2b, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A RESPIRATORY SYNCYTIAL VIRUS (RSV) VACCINE WHEN ADMINISTERED CONCOMITANTLY WITH TETANUS, DIPHTHERIA, AND ACELLULAR PERTUSSIS VACCINE (TDAP) IN HEALTHY NONPREGNANT WOMEN 18 THROUGH 49 YEARS OF AGE
Brief Title: A STUDY OF A RSV VACCINE WHEN GIVEN TOGETHER WITH TDAP IN HEALTHY NONPREGNANT WOMEN AGED BETWEEN 18 TO 49 YEARS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671004
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory tract infection; Respiratory Syncytial Virus; RSV; Tdap; Tetanus; Diphtheria; Acellular Pertussis; Vaccine
MeSH Terms: conditions — Respiratory Tract Infections; Tetanus; Diphtheria | interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an observer-blinded study. Study staff dispensing and administering the vaccine will be unblinded, but the participant and all other study personnel, including the principal investigator, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Lower RSV vaccine dose and Tdap (Experimental): Lower RSV vaccine dose and Tdap
  Interventions: Biological: RSV Vaccine; Biological: Tdap
- Lower RSV vaccine dose and Placebo (Experimental): Lower RSV vaccine dose and Placebo
  Interventions: Biological: RSV Vaccine; Biological: Placebo
- Higher RSV vaccine dose with Aluminum Hydroxide and Tdap (Experimental): Higher RSV vaccine dose with Aluminum Hydroxide and Tdap
  Interventions: Biological: RSV Vaccine; Biological: Tdap
- Higher RSV vaccine dose with Aluminum Hydroxide and Placebo (Experimental): Higher RSV vaccine dose with Aluminum Hydroxide and Placebo
  Interventions: Biological: RSV Vaccine; Biological: Placebo
- Placebo and Tdap (Placebo Comparator): Normal saline solution for injection (0.9% sodium chloride injection) and Tdap
  Interventions: Biological: Tdap; Biological: Placebo

INTERVENTIONS:
Biological: RSV Vaccine — RSV vaccine
  Arms: Higher RSV vaccine dose with Aluminum Hydroxide and Placebo; Higher RSV vaccine dose with Aluminum Hydroxide and Tdap; Lower RSV vaccine dose and Placebo; Lower RSV vaccine dose and Tdap
Biological: Tdap — Tetanus, Diphtheria, and Acellular Pertussis Vaccine
  Arms: Higher RSV vaccine dose with Aluminum Hydroxide and Tdap; Lower RSV vaccine dose and Tdap; Placebo and Tdap
Biological: Placebo — Normal saline solution for injection (0.9% sodium chloride injection)
  Arms: Higher RSV vaccine dose with Aluminum Hydroxide and Placebo; Lower RSV vaccine dose and Placebo; Placebo and Tdap

SUMMARY:
This phase 2b study will evaluate safety, tolerability, and immunogenicity of an RSV vaccine when given together with Tdap in approximately 710 healthy nonpregnant women 18 through 49 years of age. This study will evaluate non-inferiority of RSV vaccine when given with Tdap and vice-versa.

DETAILED DESCRIPTION:
This Phase 2b study will evaluate safety, tolerability, and immunogenicity of an RSV vaccine when given together with Tdap in approximately 710 healthy nonpregnant women 18 through 49 years of age.

The participants will be equally split into 5 treatment groups: One of a possible two dose levels of RSV vaccine (the higher dose level will be formulated with an aluminum hydroxide adjuvant) with either the Tdap or Placebo, or a Tdap and placebo combination.

This study will evaluate non-inferiority of the Tdap when co-administered with RSV vaccine candidate and vice-versa by measuring participants' immune response through appropriate antibody and component levels 1 month after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ≥18 and ≤49 years of age who are of childbearing potential or not of childbearing potential. (Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.)
* Willing and able to comply with all scheduled visits, treatment plan, lifestyle considerations, and other study procedures.
* Expected to be available for the duration of the study and can be contacted by telephone during study participation.
* Body mass index (BMI) of <40 kg/m2 at the time of the consent.
* Capable of giving signed informed consent as which includes compliance with the requirements and restrictions listed within.

Exclusion Criteria:

* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the vaccines being administered in the study.
* History of latex allergy.
* Immunocompromised participants with known or suspected immunodeficiency, as determined by history, laboratory tests, and/or physical examination.
* Any contraindication to Tdap (including encephalopathies).
* History of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin dependent diabetes mellitus (type 1).
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Previous vaccination with any licensed or investigational RSV vaccine, or planned receipt of nonstudy RSV vaccine throughout the study.
* Treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before investigational product administration. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Receipt of blood/plasma products or immunoglobulin within 60 days before investigational product administration or planned receipt throughout the study.
* Current alcohol abuse, marijuana abuse, or illicit drug use.
* Vaccination within 5 years with DTaP or tetanus and diphtheria toxoids adsorbed (Td) vaccine before investigational product administration.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.
* Current febrile illness (oral temperature ≥38.0C [≥100.4F]) or other acute illness within 48 hours before investigational product administration.
* Receipt of any inactivated vaccine within 14 days and any live vaccine within 28 days before or anticipated receipt of any vaccine within the 14 days after investigational product administration.
* Receipt of short-term (<14 days) systemic corticosteroids. Investigational product administration should be delayed until systemic corticosteroid use has been discontinued for at least 28 days. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids do not require temporary delay of investigational product administration.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy, non-pregnant women 18 to 49 years of age, who are of childbearing potential or not of childbearing potential.
Enrollment: 713 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Alliance for multispecialty research, Wichita, Kansas
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - Benchmark Research, Austin, Texas
  - Ventavia Research Group, Fort Worth, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc / Jordan River Family Medicine, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Peterson JT, Zareba AM, Fitz-Patrick D, Essink BJ, Scott DA, Swanson KA, Chelani D, Radley D, Cooper D, Jansen KU, Dormitzer PR, Gruber WC, Gurtman A. Safety and Immunogenicity of a Respiratory Syncytial Virus Prefusion F Vaccine When Coadministered With a Tetanus, Diphtheria, and Acellular Pertussis Vaccine. J Infect Dis. 2022 Jun 15;225(12):2077-2086. doi: 10.1093/infdis/jiab505. PMID 34637519
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671004

RESULTS

PARTICIPANT FLOW:
Groups:
- Respiratory Syncytial Virus (RSV) Vaccine 120 Microgram (mcg) With Placebo: Participants received 0.5 milliliter (mL), intramuscular injections of RSV vaccine 120 mcg (reconstituted with sterile water for injection) along with matching placebo (normal saline) on Day 1. Participants were followed up to 1 month after vaccination.
- RSV Vaccine 120 mcg With Tdap: Participants received 0.5 mL, intramuscular injections of RSV vaccine 120 mcg (reconstituted with sterile water for injection) along with tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine adsorbed (Tdap) on Day 1. Participants were followed up to 1 month after vaccination.
- RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo: Participants received 0.5 mL, intramuscular injections of RSV vaccine 240 mcg with aluminum hydroxide with matching placebo (normal saline) on Day 1. Participants were followed up to 1 month after vaccination.
- RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap: Participants received 0.5 mL, intramuscular injections of RSV vaccine 240 mcg with aluminum hydroxide with Tdap on Day 1. Participants were followed up to 1 month after vaccination.
- Placebo/Tdap: Participants received 0.5 mL, intramuscular injection of matching placebo to RSV vaccine and Tdap on Day 1. Participants were followed up to 1 month after vaccination.
Period: Overall Study
Arm/Group | Respiratory Syncytial Virus (RSV) Vaccine 120 Microgram (mcg) With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Started | 143 | 143 | 143 | 143 | 141
Treated | 141 | 141 | 143 | 143 | 141
Safety Population (Safety analysis set included all randomized participants who received investigational product. Participants were analyzed according to the investigational product they actually received.) | 141 | 141 | 142 (1 participant randomized to this arm received RSV vaccine 240 mcg with aluminum hydroxide withTdap) | 144 (1 participant of this arm actually received RSV vaccine 240 mcg with aluminum hydroxide with Tdap) | 141
Completed | 140 | 139 | 140 | 140 | 136
Not Completed | 3 | 4 | 3 | 3 | 5
Not completed — Lost to Follow-up | 1 | 2 | 3 | 3 | 5
Not completed — Randomized but not treated | 2 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received investigational product. Participants were analyzed according to the investigational product they actually received.
Groups:
- RSV Vaccine 120 mcg With Placebo: Participants received 0.5 mL, intramuscular injections of RSV vaccine 120 mcg (reconstituted with sterile water for injection) along with matching placebo (normal saline) on Day 1. Participants were followed up to 1 month after vaccination.
- RSV Vaccine 120 mcg With Tdap: Participants received 0.5 mL, intramuscular injections of RSV vaccine 120 mcg (reconstituted with sterile water for injection) along with Tdap on Day 1. Participants were followed up to 1 month after vaccination.
- Total: Total of all reporting groups
Arm/Group | RSV Vaccine 120 mcg With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap | Total
Number analyzed (Participants) | 141 | 141 | 142 | 144 | 141 | 709
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (9.2) | 35.7 (8.7) | 36.0 (8.3) | 36.1 (9.1) | 34.4 (9.2) | 35.6 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 141 | 142 | 144 | 141 | 709
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 16 | 23 | 19 | 16 | 97
  Not Hispanic or Latino | 116 | 125 | 119 | 124 | 125 | 609
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 0 | 1 | 4
  Asian | 12 | 9 | 10 | 5 | 5 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 1 | 0 | 4
  Black or African American | 29 | 28 | 25 | 29 | 38 | 149
  White | 100 | 98 | 101 | 107 | 97 | 503
  More than one race | 0 | 2 | 3 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Anti-Tetanus Toxoid (TTd) Antibody Concentrations of Greater Than or Equal to (>=) 0.1 International Units Per Milliliter (IU/mL) at 1 Month After Vaccination
Description: Percentage of participants achieving Anti-TTd antibody concentrations of >= 0.1 IU/mL at 1 month after vaccination were reported. The lower limit of quantitation (LLOQ) values for Anti-TTd was 0.05 IU/mL. Assay results below the LLOQ were set to 0.5*LLOQ. Data for this outcome measure was planned to be collected and analyzed only for combined population of participants reported under two RSV vaccine arms: (RSV vaccine 120 mcg with Tdap and RSV vaccine 240 mcg with aluminum hydroxide/Tdap) along with placebo/Tdap arm and not planned to be collected and analyzed for two RSV vaccine arms: (RSV vaccine 120 mcg with placebo and RSV vaccine 240 mcg with aluminum hydroxide with placebo), as pre-specified in protocol.
Time Frame: 1 month after vaccination
Population: Evaluable immunogenicity population(EIP): participants who were eligible, received all doses of investigational product to which they were randomized, had blood drawn for assay testing within specified time frame for 1 month after vaccination, had >=1 valid, determinate assay result at 1-month-postvaccination visit and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSV Vaccine With Aluminum Hydroxide With Tdap: This arm included all participants who received 0.5 mL intramuscular injection of either RSV vaccine 120 mcg (reconstituted with sterile water for injection) along with Tdap or RSV vaccine 240 mcg with aluminum hydroxide with Tdap on Day 1. Participants were followed up to 1 month after vaccination.
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 272 | 134
Percentage of participants | 100 [98.7 to 100.0] | 100 [97.3 to 100.0]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs Placebo/Tdap; Difference in percentage; Test type: Superiority; Difference in proportions = 0.0, 95% CI 2-sided [-1.4 to 2.8]

2. Primary Outcome: Percentage of Participants Achieving Anti-Diphtheria Toxoid (DTd) Antibody Concentrations of >= 0.1 IU/mL at 1 Month After Vaccination
Description: Percentage of participants achieving Anti-DTd antibody concentrations of >= 0.1 IU/mL at 1 month after vaccination were reported. The LLOQ values for Anti- DTd= 0.037 IU/mL. Assay results below the LLOQ were set to 0.5*LLOQ. Data for this outcome measure was planned to be collected and analyzed only for combined population of participants reported under two RSV vaccine arms: (RSV vaccine 120 mcg with Tdap and RSV vaccine 240 mcg with aluminum hydroxide/Tdap) along with placebo/Tdap arm and not planned to be collected and analyzed for two RSV vaccine arms: (RSV vaccine 120 mcg with placebo and RSV vaccine 240 mcg with aluminum hydroxide with placebo), as pre-specified in protocol.
Time Frame: 1 month after vaccination
Population: EIP: participants who were eligible, received all doses of investigational product to which they were randomized, have blood drawn for assay testing within the specified time frame for 1 month after vaccination, had at least 1 valid and determinate assay result at the 1-month-postvaccination visit and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 272 | 134
Percentage of participants | 97.4 [94.8 to 99.0] | 99.3 [95.9 to 100.0]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs Placebo/Tdap; Difference in percentage; Test type: Superiority; Difference in proportions = -1.8, 95% CI 2-sided [-4.6 to 1.7]

3. Primary Outcome: Geometric Mean Concentration (GMC) and Geometric Mean Ratio (GMR) of Anti-Pertussis Antibodies 1 Month After Vaccination
Description: GMCs of anti-pertussis components: anti pertussis (anti-PT) toxin, anti filamentous hemagglutinin (FHA) and anti- pertactin (PRN) was measured and reported in descriptive section. LLOQ values for each component was: Anti-PT=0.9 endotoxin units per milliliter (EU/mL), Anti-FHA=2.9 EU/mL, and Anti-PRN=3.0 EU/mL. Assay results below LLOQ were set to 0.5*LLOQ. Descriptive data for this outcome measure was planned to be collected and analyzed only for combined population of participants reported under two RSV vaccine arms: (RSV vaccine 120 mcg with Tdap and RSV vaccine 240 mcg with aluminum hydroxide/Tdap) along with placebo/Tdap arm and not planned to be collected and analyzed for two RSV vaccine arms: (RSV vaccine 120 mcg with placebo and RSV vaccine 240 mcg with aluminum hydroxide with placebo), as pre-specified in protocol. GMRs were reported in statistical analysis section and calculated by dividing GMC of RSV vaccine with aluminum hydroxide with Tdap arm by GMC of placebo/Tdap arm.
Time Frame: 1 month after vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Endotoxin unit per milliliter (EU/mL)
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 272 | 134
Endotoxin unit per milliliter (EU/mL)
  Anti-PT | 36.59 [33.10 to 40.46] | 45.90 [37.43 to 56.29]
  Anti-FHA | 113.30 [104.13 to 123.28] | 191.33 [164.46 to 222.59]
  Anti-PRN | 154.13 [135.98 to 174.70] | 257.05 [211.55 to 312.34]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs Placebo/Tdap; Anti-PT: Ratio of geometric mean was calculated by dividing the GMC of RSV vaccine with aluminum hydroxide with Tdap arm by GMC of placebo/Tdap arm; Test type: Superiority; Ratio of Geometric Mean = 0.80, 95% CI 2-sided [0.64 to 1.00]
Statistical Analysis 2: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs Placebo/Tdap; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Ratio of Geometric Mean = 0.59, 95% CI 2-sided [0.50 to 0.70]
Statistical Analysis 3: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs Placebo/Tdap; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Ratio of Geometric Mean = 0.60, 95% CI 2-sided [0.48 to 0.76]

4. Primary Outcome: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Respiratory Syncytial Virus Subgroup A (RSV A) Neutralizing Antibodies 1 Month After Vaccination Using 2.0 Fold Margin
Description: Assay results below the LLOQ were set to 0.5*LLOQ. Titers were expressed in terms of 1/dilution. Descriptive data for this outcome measure was planned to be collected and analyzed for combined population of participants reported under two RSV and Tdap vaccine arms: (RSV vaccine 120 mcg with Tdap and RSV vaccine 240 mcg with aluminum hydroxide/Tdap) and two RSV and placebo arm: (RSV vaccine 120 mcg with placebo and RSV vaccine 240 mcg with aluminum hydroxide with placebo) and not planned to be collected and analyzed for Placebo/Tdap arm, as pre-specified in protocol. GMRs were reported in statistical analysis section and calculated by dividing GMT of RSV vaccine with aluminum hydroxide with Tdap arm by GMT of RSV vaccine with aluminum hydroxide with placebo arm.
Time Frame: 1 month after vaccination
Population: EIP: participants who were eligible, received all doses of investigational product to which they were randomized, have blood drawn for assay testing within the specified time frame for 1 month after vaccination, had at least 1 valid and determinate assay result at the 1-month-postvaccination visit and had no major protocol violations. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- RSV Vaccine With Aluminum Hydroxide With Placebo: This arm included all participants who received 0.5 mL intramuscular injection of either RSV vaccine 120 mcg (reconstituted with sterile water for injection) along with matching placebo or RSV vaccine 240 mcg with aluminum hydroxide with matching placebo on Day 1. Participants were followed up to 1 month after vaccination.
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | RSV Vaccine With Aluminum Hydroxide With Placebo
Number analyzed (Participants) | 272 | 270
Titer | 22339.0 [20362.3 to 24507.6] | 22980.1 [20371.3 to 25922.9]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs RSV Vaccine With Aluminum Hydroxide With Placebo; 2.0-fold margin (related to primary objective): primary objective was demonstrated if the lower limit of 95% confidence interval (CI) from the ratio of titers with 50 percent cut off from two treatment groups greater than (>) 0.5; Test type: Superiority; Ratio of Geometric Mean = 0.97, 95% CI 2-sided [0.84 to 1.13] — Ratio of geometric mean was calculated by dividing GMT of RSV vaccine with aluminum hydroxide with Tdap arm by GMT of RSV vaccine with aluminum hydroxide with placebo arm

5. Primary Outcome: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Respiratory Syncytial Virus Subgroup B (RSV B) Neutralizing Antibodies 1 Month After Vaccination Using 2.0 Fold Margin
Description: as for outcome 4
Time Frame: 1 month after vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | RSV Vaccine With Aluminum Hydroxide With Placebo
Number analyzed (Participants) | 272 | 271
Titer | 21509.7 [19279.4 to 23997.9] | 22486.0 [19696.2 to 25671.0]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs RSV Vaccine With Aluminum Hydroxide With Placebo; 2.0-fold margin (related to primary objective): primary objective was demonstrated if the lower limit of 95% CI from the ratio of titers with 50 percent cut off from two treatment groups > 0.5; Test type: Superiority; Ratio of Geometric Mean = 0.96, 95% CI 2-sided [0.81 to 1.14] — [estimate comment as in outcome 4, analysis 1]

6. Primary Outcome: Percentage of Participants With Prespecified Local Reactions Within 7 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity.
Time Frame: Within 7 days after vaccination
Population: Safety analysis set included all randomized participants who received investigational product. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine 120 mcg With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 141 | 141 | 141 | 143 | 139
Percentage of participants
  Pain at injection site: mild | 33.3 [25.6 to 41.8] | 34.0 [26.3 to 42.5] | 46.1 [37.7 to 54.7] | 46.9 [38.5 to 55.4] | 21.6 [15.1 to 29.4]
  Pain at injection site: moderate | 7.1 [3.5 to 12.7] | 9.9 [5.5 to 16.1] | 19.9 [13.6 to 27.4] | 15.4 [9.9 to 22.4] | 4.3 [1.6 to 9.2]
  Pain at injection site: severe | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.9] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Redness: mild | 6.4 [3.0 to 11.8] | 3.5 [1.2 to 8.1] | 4.3 [1.6 to 9.0] | 2.8 [0.8 to 7.0] | 0.7 [0.0 to 3.9]
  Redness: moderate | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.9] | 2.8 [0.8 to 7.0] | 0 [0.0 to 2.6]
  Redness: severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Swelling: mild | 4.3 [1.6 to 9.0] | 4.3 [1.6 to 9.0] | 2.1 [0.4 to 6.1] | 3.5 [1.1 to 8.0] | 0.7 [0.0 to 3.9]
  Swelling: moderate | 2.8 [0.8 to 7.1] | 1.4 [0.2 to 5.0] | 2.1 [0.4 to 6.1] | 3.5 [1.1 to 8.0] | 0.7 [0.0 to 3.9]
  Swelling: severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]

7. Primary Outcome: Percentage of Participants With Prespecified Systemic Reactions Within 7 Days After Vaccination
Description: Systemic reactions included fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever was categorized as: >=38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
Time Frame: Within 7 days after vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine 120 mcg With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 141 | 141 | 141 | 143 | 139
Percentage of participants
  Fever: >=38.0 degree C | 7.8 [4.0 to 13.5] | 6.4 [3.0 to 11.8] | 6.4 [3.0 to 11.8] | 7.7 [3.9 to 13.3] | 5.0 [2.0 to 10.1]
  Fever: mild | 4.3 [1.6 to 9.0] | 3.5 [1.2 to 8.1] | 5.7 [2.5 to 10.9] | 2.8 [0.8 to 7.0] | 3.6 [1.2 to 8.2]
  Fever: moderate | 2.1 [0.4 to 6.1] | 1.4 [0.2 to 5.0] | 0.7 [0.0 to 3.9] | 3.5 [1.1 to 8.0] | 0.7 [0.0 to 3.9]
  Fever: severe | 1.4 [0.2 to 5.0] | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 1.4 [0.2 to 5.0] | 0 [0.0 to 2.6]
  Fever: Grade 4 | 0 [0.0 to 2.6] | 1.4 [0.2 to 5.0] | 0 [0.0 to 2.6] | 0 [0.0 to 2.5] | 0.7 [0.0 to 3.9]
  Fatigue: mild | 20.6 [14.2 to 28.2] | 24.1 [17.3 to 32.0] | 21.3 [14.8 to 29.0] | 23.1 [16.4 to 30.9] | 26.6 [19.5 to 34.8]
  Fatigue: moderate | 19.1 [13.0 to 26.6] | 22.0 [15.5 to 29.7] | 22.7 [16.1 to 30.5] | 22.4 [15.8 to 30.1] | 17.3 [11.4 to 24.6]
  Fatigue: severe | 2.8 [0.8 to 7.1] | 2.1 [0.4 to 6.1] | 0.7 [0.0 to 3.9] | 1.4 [0.2 to 5.0] | 0 [0.0 to 2.6]
  Headache: mild | 17.0 [11.2 to 24.3] | 20.6 [14.2 to 28.2] | 27.0 [19.8 to 35.1] | 24.5 [17.7 to 32.4] | 20.1 [13.8 to 27.8]
  Headache: moderate | 16.3 [10.6 to 23.5] | 19.9 [13.6 to 27.4] | 17.7 [11.8 to 25.1] | 14.7 [9.3 to 21.6] | 15.8 [10.2 to 23.0]
  Headache: severe | 2.1 [0.4 to 6.1] | 1.4 [0.2 to 5.0] | 1.4 [0.2 to 5.0] | 2.1 [0.4 to 6.0] | 0.7 [0.0 to 3.9]
  Nausea: mild | 9.9 [5.5 to 16.1] | 11.3 [6.6 to 17.8] | 9.9 [5.5 to 16.1] | 12.6 [7.6 to 19.2] | 13.7 [8.4 to 20.5]
  Nausea: moderate | 12.1 [7.2 to 18.6] | 5.7 [2.5 to 10.9] | 5.7 [2.5 to 10.9] | 7.0 [3.4 to 12.5] | 7.9 [4.0 to 13.7]
  Nausea: severe | 0.7 [0.0 to 3.9] | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Muscle pain: mild | 19.1 [13.0 to 26.6] | 33.3 [25.6 to 41.8] | 31.9 [24.3 to 40.3] | 30.1 [22.7 to 38.3] | 23.0 [16.3 to 30.9]
  Muscle pain: moderate | 15.6 [10.0 to 22.7] | 15.6 [10.0 to 22.7] | 15.6 [10.0 to 22.7] | 22.4 [15.8 to 30.1] | 11.5 [6.7 to 18.0]
  Muscle pain: severe | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.8] | 0 [0.0 to 2.6]
  Joint pain: mild | 7.8 [4.0 to 13.5] | 11.3 [6.6 to 17.8] | 9.2 [5.0 to 15.3] | 9.1 [4.9 to 15.0] | 4.3 [1.6 to 9.2]
  Joint pain: moderate | 7.1 [3.5 to 12.7] | 6.4 [3.0 to 11.8] | 7.8 [4.0 to 13.5] | 8.4 [4.4 to 14.2] | 7.2 [3.5 to 12.8]
  Joint pain: severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Vomiting: mild | 3.5 [1.2 to 8.1] | 4.3 [1.6 to 9.0] | 0.7 [0.0 to 3.9] | 2.1 [0.4 to 6.0] | 2.2 [0.4 to 6.2]
  Vomiting: moderate | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9] | 0.7 [0.0 to 3.9] | 0 [0.0 to 2.5] | 2.2 [0.4 to 6.2]
  Vomiting: severe | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]
  Diarrhea: mild | 12.1 [7.2 to 18.6] | 13.5 [8.3 to 20.2] | 9.2 [5.0 to 15.3] | 10.5 [6.0 to 16.7] | 10.1 [5.6 to 16.3]
  Diarrhea: moderate | 3.5 [1.2 to 8.1] | 5.0 [2.0 to 10.0] | 1.4 [0.2 to 5.0] | 6.3 [2.9 to 11.6] | 5.0 [2.0 to 10.1]
  Diarrhea: severe | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9] | 1.4 [0.2 to 5.0] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]

8. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Within 1 month after vaccination (up to 35 days)
Population: Safety analysis set included all randomized participants who received investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine 120 mcg With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 141 | 141 | 142 | 144 | 141
Percentage of participants | 5.7 [2.5 to 10.9] | 7.8 [4.0 to 13.5] | 5.6 [2.5 to 10.8] | 10.4 [5.9 to 16.6] | 9.2 [5.0 to 15.3]

9. Primary Outcome: Percentage of Participants With Medically Attended Adverse Events (MAE) and Serious Adverse Events (SAE)
Description: An medically attended adverse events (MAE) was defined as a non-serious AE that results in an evaluation at a medical facility. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Within 1 month after vaccination (up to 35 days)
Population: Safety analysis set included all randomized participants who received investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine 120 mcg With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 141 | 141 | 142 | 144 | 141
Percentage of participants
  SAE | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 0.7 [0.0 to 3.9] | 0 [0.0 to 2.5] | 0 [0.0 to 2.6]
  MAE | 1.4 [0.2 to 5.0] | 0 [0.0 to 2.6] | 0 [0.0 to 2.6] | 1.4 [0.2 to 4.9] | 2.1 [0.4 to 6.1]

10. Secondary Outcome: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Respiratory Syncytial Virus Subgroup A (RSV A) Neutralizing Antibodies 1 Month After Vaccination Using 1.5 Fold Margin
Description: as for outcome 4
Time Frame: 1 month after vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | RSV Vaccine With Aluminum Hydroxide With Placebo
Number analyzed (Participants) | 272 | 270
Titer | 22339.0 [20362.3 to 24507.6] | 22980.1 [20371.3 to 25922.9]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs RSV Vaccine With Aluminum Hydroxide With Placebo; 1.5-fold margin (related to secondary objective): secondary objective was demonstrated if the lower limit of 95% CI from the ratio of titers with 50 percent cut off from two treatment groups > 0.67; Test type: Superiority; Ratio of Geometric Mean = 0.97, 95% CI 2-sided [0.84 to 1.13] — [estimate comment as in outcome 4, analysis 1]

11. Secondary Outcome: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Respiratory Syncytial Virus Subgroup B (RSV B) Neutralizing Antibodies 1 Month After Vaccination Using 1.5 Fold Margin
Description: as for outcome 4
Time Frame: 1 month after vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | RSV Vaccine With Aluminum Hydroxide With Placebo
Number analyzed (Participants) | 272 | 271
Titer | 21509.7 [19279.4 to 23997.9] | 22486.0 [19696.2 to 25671.0]
Statistical Analysis 1: Comparison: RSV Vaccine With Aluminum Hydroxide With Tdap vs RSV Vaccine With Aluminum Hydroxide With Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; Ratio of Geometric Mean = 0.96, 95% CI 2-sided [0.81 to 1.14] — [estimate comment as in outcome 4, analysis 1]

12. Other Pre Specified Outcome: Percentage of Participants Achieving Anti-TTd Antibody Concentrations of >= 0.1 IU/mL Before Vaccination
Description: Percentage of participants achieving Anti-TTd antibody concentrations of >= 0.1 IU/mL 1 month before vaccination were reported. The LLOQ values for Anti-TTd = 0.05 IU/mL. Assay results below the LLOQ were set to 0.5*LLOQ. Data for this outcome measure was not planned to be collected and analyzed for RSV 120 mcg with placebo arm and RSV 240 mcg with aluminum hydroxide/placebo arm.
Time Frame: Before vaccination on Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 135 | 137 | 134
Percentage of participants | 97.8 [93.6 to 99.5] | 96.4 [91.7 to 98.8] | 99.3 [95.9 to 100.0]

13. Other Pre Specified Outcome: Percentage of Participants Achieving Anti- DTd Antibody Concentrations of >= 0.1 IU/mL Before Vaccination
Description: Percentage of participants achieving Anti-DTd antibody concentrations of >= 0.1 IU/mL before vaccination were reported. The LLOQ values for Anti-DTd= 0.037 IU/mL. Assay results below the LLOQ were set to 0.5*LLOQ. Data for this outcome measure was not planned to be collected and analyzed for RSV 120 mcg with placebo arm and RSV 240 mcg with aluminum hydroxide/placebo arm.
Time Frame: Before vaccination on Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
Number analyzed (Participants) | 135 | 137 | 134
Percentage of participants | 83.0 [75.5 to 88.9] | 78.8 [71.0 to 85.3] | 82.1 [74.5 to 88.2]

14. Other Pre Specified Outcome: Geometric Mean Titer (GMT) of Respiratory Syncytial Virus Subgroup A (RSV A) Neutralizing Antibodies Before Vaccination
Description: Assay results below the LLOQ were set to 0.5*LLOQ. Titers were expressed in terms of 1/dilution. Data for this outcome measure was planned to be collected and analyzed for combined population of participants reported under two RSV and Tdap vaccine arms: (RSV vaccine 120 mcg with Tdap and RSV vaccine 240 mcg with aluminum hydroxide/Tdap) and two RSV and placebo arm: (RSV vaccine 120 mcg with placebo and RSV vaccine 240 mcg with aluminum hydroxide with placebo) and not planned to be collected and analyzed for Placebo/Tdap arm, as pre-specified in protocol.
Time Frame: Before vaccination on Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | RSV Vaccine With Aluminum Hydroxide With Placebo
Number analyzed (Participants) | 272 | 271
Titer | 1582.6 [1450.3 to 1726.9] | 1560.6 [1419.4 to 1715.8]

15. Other Pre Specified Outcome: Geometric Mean Titer (GMT) of Respiratory Syncytial Virus Subgroup B (RSV B) Neutralizing Antibodies Before Vaccination
Description: as for outcome 14
Time Frame: Before vaccination on Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | RSV Vaccine With Aluminum Hydroxide With Tdap | RSV Vaccine With Aluminum Hydroxide With Placebo
Number analyzed (Participants) | 272 | 271
Titer | 1470.2 [1343.6 to 1608.7] | 1417.3 [1284.8 to 1563.5]

ADVERSE EVENTS:
Time Frame: Local reactions and systematic reactions: within 7 days after vaccination. AEs: Baseline up to 35 days
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | RSV Vaccine 120 mcg With Placebo | RSV Vaccine 120 mcg With Tdap | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap | Placebo/Tdap
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/141 | 0/142 | 0/144 | 0/141
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/141 | 1/142 | 0/144 | 0/141
Other Adverse Events (participants affected / at risk) | 103/141 | 114/141 | 118/142 | 119/144 | 106/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSV Vaccine 120 mcg With Placebo (N=141) | RSV Vaccine 120 mcg With Tdap (N=141) | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo (N=142) | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap (N=144) | Placebo/Tdap (N=141)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RSV Vaccine 120 mcg With Placebo (N=141) | RSV Vaccine 120 mcg With Tdap (N=141) | RSV Vaccine 240 mcg With Aluminum Hydroxide With Placebo (N=142) | RSV Vaccine 240 mcg With Aluminum Hydroxide With Tdap (N=144) | Placebo/Tdap (N=141)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 22 | 27 | 17 | 24 | 21
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 32 | 24 | 22 | 28 | 30
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 7 | 3 | 3 | 6
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 60 | 68 | 63 | 67 | 61
Fatigue (General disorders) | 0 | 3 | 0 | 1 | 1
Injection site erythema (General disorders) | 10 | 6 | 7 | 8 | 1
Injection site pain (General disorders) | 57 | 63 | 94 | 89 | 36
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 10 | 8 | 6 | 10 | 2
Pyrexia (General disorders) | 11 | 9 | 9 | 11 | 7
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Venomous sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 25 | 24 | 25 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 49 | 70 | 68 | 76 | 48
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 50 | 59 | 65 | 59 | 51
Headache (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04071158/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/58/NCT04071158/SAP_001.pdf